CLINICAL TRIAL: NCT07325279
Title: A Phase 1, Open-Label, Safety, Tolerability, and Pharmacokinetic Study of Nalmefene Implants in Healthy Subjects
Brief Title: Nalmefene Implant in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ReacX Pharmaceuticals, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NI-001; 5UGDA047707-02 (Other Grant/Funding Number: NIDA)
Record Dates: First submitted 2025-12-17; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Opioid Abuse and Addiction
Keywords: nalmefene implant opioid addition
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1; 1 Implant (Active Comparator)
  Interventions: Drug: 1 Nalmefene implant
- Cohort 2; 2 Implants (Active Comparator)
  Interventions: Drug: 2 Nalmefene implants

INTERVENTIONS:
Drug: 1 Nalmefene implant — One implant
  Arms: Cohort 1; 1 Implant
Drug: 2 Nalmefene implants — Two Implants
  Arms: Cohort 2; 2 Implants

SUMMARY:
The goal of this clinical trial is to learn how safe either one or two nalmefene implants are after remaining implanted for 4 or 12 weeks.

Additionally the pharmacokinetics (PK), how fast the drug is absorbed into the body and how long it remains in the body, will also be studies.

The data collected in this healthy volunteer study will inform the Sponsor on how best to proceed with future trials in the intended patient population.

DETAILED DESCRIPTION:
This is a single center, Phase 1, open-label, safety, tolerability, and PK study designed to compare one (1) or two (2) nalmefene implants in healthy subjects.

The study will include a screening period from Day -28 to Day -2, where subjects will be evaluated according to the Inclusion/Exclusion Criteria. Enrollment will be initially restricted to Cohort 1 (1 implant) until the Safety Review Committee (SRC) completes an evaluation of the safety data, of at least 5 subjects, through the Week 4 Visit. The SRC will then advise the Sponsor as to whether to open enrollment to Cohort 2 (2 implants).

Including screening, the first 8 subjects will be enrolled into Cohort 1 Subgroup 1 and will be seen for 16 visits over a period of up to 18 weeks. This includes a total of up to 8 nights of inpatient stay during that period. Eligible subjects will be admitted to the clinical site on Day -1 and implant insertion will occur on Day 1. Subjects will be confined until completion of the assessments on Day 2. Subjects will return to the clinical site for outpatient visits on Days 3 and 4, and Weeks 1, 2, 3, 4, 6, 8, and 10. Subjects will be admitted again two days prior to the Week 12/End of Treatment for an implant removal visit and will be discharged after the final blood sample is collected 72 hours after implant removal. Subjects will return to the clinical site for follow-up visits on Week 13 and Week 14 (1 and 2 week(s) following implant removal procedure) for removal of sutures (if any) and safety evaluations.

Including screening, subjects enrolled into Cohort 1 Subgroup 2 and Cohort 2 will be seen for approximately 22 visits over a period of up to 30 weeks. This includes a total of 8 nights of inpatient stay during that period. Eligible subjects will be admitted to the clinical site on Day -1 and implant insertion will occur on Day 1. Subjects will be confined until completion of the assessments on Day 2. Subjects will return to the clinical site for outpatient visits on Days 3 and 4, and Weeks 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, and 22. Subjects will be admitted again on the day prior to the Week 24/EOT implant removal visit and will be discharged after the final blood sample is collected 72 hours after implant removal. Subjects will return to the clinical site for follow-up visits on Week 25 and Week 26 (1 and 2 week(s) following implant removal procedure) for removal of sutures (if any) and safety evaluations.

ELIGIBILITY:
Inclusion Criteria:

- Subjects must meet all of the following criteria to be included in the study:

1. Male or female, non-smoker, ≥18 and ≤55 years of age, with body mass index (BMI) >18.5 and <35.0 kg/m2 and body weight ≥50.0 kg for males and ≥45.0 kg for females.
2. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 4 weeks prior to implant insertion.
   2. the absence of clinically significant history of dermatologic, neurological, musculoskeletal, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
3. Female subjects of non-childbearing potential must be:

   1. post-menopausal with confirmation by documented follicle-stimulating hormone (FSH) test; or
   2. surgically sterile .
4. Female subjects of childbearing potential who are sexually active with a non-sterile male partner must be willing to use an acceptable contraceptive methods throughout the study and for 30 days after the implant is removed:
5. Male subjects who are not vasectomized for at least 3 months prior to implant insertion and who are sexually active with a female partner of childbearing potential must be willing to use an acceptable contraceptive methods from implant insertion and for 30 days after the implant is removed:

6 Able to understand the study procedures and provide signed informed consent to participate in the study.

Exclusion Criteria:

* Subjects to whom any of the following applies will be excluded from the study:

  1. Any clinically significant abnormal finding at physical examination at screening.
  2. Clinically significant history of or current evidence of suicidal ideation or active suicidal behavior as based on the C-SSRS.
  3. Clinically significant history or current evidence of depression as based on the MADRS.
  4. Clinically significant abnormal laboratory test results or positive serology test results for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antigen and antibody at screening.
  5. Positive pregnancy test or lactating female subject.
  6. Positive urine drug screen, urine cotinine test, or alcohol breath test.
  7. Known medically significant intolerance or allergic reactions to nalmefene or to ethylene vinyl acetate
  8. Hypersensitivity to lidocaine or other local anesthetics of the amide type, epinephrine, antiseptic solution
  9. Clinically significant ECG abnormalities or vital signs abnormalities
  10. History of drug use within 1 year prior to screening or recreational use of marijuana within 1 month
  11. History of alcohol abuse within 1 year prior to screening
  12. Use of medications for the timeframes specified below:

      1. depot injection or implant within 3 months prior to implant insertion;
      2. any drug known to induce hepatic drug metabolism within 30 days prior to implant insertion;
      3. prescription medications within 14 days prior to implant insertion;
      4. any vaccine within 14 days prior to implant insertion;
      5. over-the-counter medications and natural health products within 7 days prior to implant insertion
  13. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to implant insertion,
  14. Donation of plasma within 7 days prior to dosing or donation or
  15. Intolerant to venipuncture and/or have difficulty with venous access.
  16. History of wound healing problems.
  17. Lymphedema, scarring, or tattoos on his/her inner upper arms within 2 months prior to screening or a history of keloid scarring.
  18. Any dermatologic disorder, including cancer, that precludes the safety of the implant
  19. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-07 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) after implantation with 1 or 2 nalmefene implants. | Day 1 up to Week 12 or Week 24
Columbia-Suicide Severity Rating Scale (C-SSRS) | Day 1 and Day 2
  Questionnaire
Montgomery-Asberg Depression Rating Scale (MADRS) | Day 1 and Day 2
  Questionnaire

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of nalmefene after implantation with 1 or 2 nalmefene implants. | Day 1, 2, 3, 4, Weeks 2, 3, 4, 6, 8, 10, 12, 13, 14, 16, 18, 20, 22, 24, 25, 26
  PK blood sample
Area under the concentration curve (AUC) after implantation with 1 or 2 nalmefene implants | Day 1, 2, 3, 4, Weeks 2, 3, 4, 6, 8, 10, 12, 13, 14, 16, 18, 20, 22, 24, 25, 26
  PK blood sample
Plasma concertation of nalmefene after implantation with 1 or 2 nalmefene implants | Day 1, 2, 3, 4, Weeks 2, 3, 4, 6, 8, 10, 12, 13, 14, 16, 18, 20, 22, 24, 25, 26
  PK blood sample

IPD SHARING:
Plan to Share IPD: No